CLINICAL TRIAL: NCT05875727
Title: A PHASE 3, SINGLE-ARM, MULTICENTER TRIAL TO DESCRIBE THE SAFETY AND IMMUNOGENICITY OF A 20-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN PNEUMOCOCCAL VACCINE-NAÏVE ADULTS ≥18 YEARS OF AGE IN INDIA
Brief Title: A Study to Learn About the Safety and Immune Response of 20vPnC in Adults in India.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B7471010
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Intervention Model Description: Participants will be assigned into 2 cohorts by age: 18 to 49 years of age and ≥50 years of age.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 20-valent pneumococcal conjugate vaccine (Experimental): Pneumococcal conjugate vaccine (20vPnC)
  Interventions: Biological: 20-valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 20-valent pneumococcal conjugate vaccine — One dose of 20vPnC will be administered intramuscularly.

SUMMARY:
The purpose of this study is to learn about the safety and immune response of 20vPnC in adults in India.

This study is seeking participants who:

* are generally healthy adults of 18 years or older.
* have not received pneumococcal vaccine.

The study will have 2 groups based on age. One group will have particpants between 18 to 49 years of age. The other group will have participants of 50 years or older.

Participants will take part in the study for about one month which includes two visits to the study clinic. Participants will receive a single dose of study vaccine (20vPnC) into the arm at visit 1 and will come to study site for a follow-up visit after about a month.

The study team will ask questions about the participant's health and blood samples will be taken in a subset of participants during the visits.

ELIGIBILITY:
Inclusion Criteria:

- Generally healthy participants ≥18 years of age at the time of consent.

Exclusion Criteria:

* History of severe adverse reaction associated with a vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of 20vPnC, or to any other diphtheria toxoid-containing vaccine.
* Known or suspected immune deficiency or suppression.
* Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Previous vaccination with any pneumococcal vaccine, or planned receipt of any pneumococcal vaccine through study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2023-08-16 (Actual); Primary Completion 2023-10-02 (Actual); Study Completion 2023-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- India (8):
  - Nirmal Hospital Pvt Ltd., Surat, Gujarat
  - BGS Global Institute of Medical Sciences (BGSGIMS), Bangalore, Karnataka
  - RajaRajeswari Medical College and Hospital, Bangalore, Karnataka
  - RajaRajeswari Medical College and Hospital, Bengaluru, Karnataka
  - Bharati Vidyapeeth (Deemed to be University) Medical College Hospital & Research Centre, Pune, Maharashtra
  - Aakash Healthcare Private Limited, New Delhi, National Capital Territory of Delhi
  - Jawahar Lal Nehru Hospital, Ajmer, Rajasthan
  - Jawahar Lal Nehru Medical College, Ajmer, Rajasthan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Giriappa B, Choraria N, Ponce P, Drozd J, Su X, Lei L, Portka M, Pai S, Anderson A, Bickham K, Watson W, McElwee K. Immunogenicity and safety of 20-valent pneumococcal conjugate vaccine in pneumococcal vaccine-naive adults >/=18 years of age in India: A phase 3 single-arm trial. Hum Vaccin Immunother. 2026 Dec;22(1):2605847. doi: 10.1080/21645515.2025.2605847. Epub 2026 Jan 7. PMID 41504209
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 405 participants signed the informed consent form. Two participants were screen failures and 3 were not assigned to receive study treatment and 400 participants received study treatment.
Groups:
- Cohort 1: 18 to 49 Years: Pneumococcal vaccine naive participants aged 18 to 49 years were administered 0.5 milliliter (mL) of 20-valent pneumococcal conjugate vaccine (20vPnC) vaccine, intramuscularly (IM) on Day 1 (Visit 1).
- Cohort 2: >=50 Years: Pneumococcal vaccine naive participants aged more than or equal to (>=)50 years were administered 0.5 mL of 20vPnC vaccine, IM on Day 1 (Visit 1).
Period: Overall Study
Arm/Group | Cohort 1: 18 to 49 Years | Cohort 2: >=50 Years
Started | 200 | 200
Completed | 200 | 200
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any study intervention and had safety data assessed after vaccination.
Groups:
- Cohort 1: 18 to 49 Years: Pneumococcal vaccine naive participants aged 18 to 49 years were administered 0.5 mL of 20vPnC vaccine, IM on Day 1 (Visit 1).
- Cohort 2: >= 50 Years: Pneumococcal vaccine naive participants aged >=50 years were administered 0.5 mL of 20vPnC vaccine, IM on Day 1 (Visit 1).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: 18 to 49 Years | Cohort 2: >= 50 Years | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.7 (8.18) | 58.8 (7.22) | 46.7 (14.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 52 | 116
  Male | 136 | 148 | 284
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 200 | 200 | 400
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 200 | 200 | 400
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Vaccination
Description: Local reactions (redness, swelling, and injection site pain) at the site of investigational product administration were recorded in electronic diary (e-diary). Redness and swelling were measured and recorded in caliper units where 1 caliper unit = 0.5 centimeter (cm). Redness and swelling were graded as mild (more than [>]2.0 to 5.0 cm), moderate (>5.0 to 10.0cm) and severe (>10.0cm). Pain at injection site was graded as mild (did not interfere with activity), moderate (interfered with activity), and severe (prevented daily activity). Exact 2-sided 95% confidence interval was based on the Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: 18 to 49 Years | Cohort 2: >= 50 Years
Number analyzed (Participants) | 200 | 200
Percentage of participants
  Redness: Any | 1.0 [0.1 to 3.6] | 1.0 [0.1 to 3.6]
  Redness: Mild | 0.0 [0.0 to 1.8] | 0.5 [0.0 to 2.8]
  Redness: Moderate | 0.5 [0.0 to 2.8] | 0.5 [0.0 to 2.8]
  Redness: Severe | 0.5 [0.0 to 2.8] | 0.0 [0.0 to 1.8]
  Swelling: Any | 1.5 [0.3 to 4.3] | 1.5 [0.3 to 4.3]
  Swelling: Mild | 0.5 [0.0 to 2.8] | 0.5 [0.0 to 2.8]
  Swelling: Moderate | 0.5 [0.0 to 2.8] | 1.0 [0.1 to 3.6]
  Swelling: Severe | 0.5 [0.0 to 2.8] | 0.0 [0.0 to 1.8]
  Pain at the injection site: Any | 43.5 [36.5 to 50.7] | 32.0 [25.6 to 38.9]
  Pain at the injection site: Mild | 33.5 [27.0 to 40.5] | 27.5 [21.4 to 34.2]
  Pain at the injection site: Moderate | 9.5 [5.8 to 14.4] | 4.0 [1.7 to 7.7]
  Pain at the injection site: Severe | 0.5 [0.0 to 2.8] | 0.5 [0.0 to 2.8]

2. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination
Description: Systemic events included: fever, fatigue, headache, joint pain and muscle pain. Fever was defined as an oral temperature of more than or equal to (>=)38.0 degree Celsius (C) and was classified as >=38.0 degree C, >=38.0 to 38.4 degree C, >38.4 to 38.9 degree C, >38.9 to 40.0 degree C and >40.0 degree C. Fatigue, headache, joint pain and muscle pain were graded as mild (did not interfere with activity), moderate (some interference with activity) and severe (prevented daily activity). Exact 2-sided 95% confidence interval was based on the Clopper and Pearson method.
Time Frame: Day 1 to Day 7 after vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: 18 to 49 Years | Cohort 2: >= 50 Years
Number analyzed (Participants) | 200 | 200
Percentage of participants
  Fever: >= 38.0 degree C | 3.0 [1.1 to 6.4] | 1.5 [0.3 to 4.3]
  Fever: >=38.0 to 38.4 degree C | 1.5 [0.3 to 4.3] | 0.5 [0.0 to 2.8]
  Fever: >38.4 to 38.9 degree C | 0 [0.0 to 1.8] | 1.0 [0.1 to 3.6]
  Fever: >38.9 to 40.0 degree C | 1.5 [0.3 to 4.3] | 0 [0.0 to 1.8]
  Fever: >40.0 degree C | 0 [0.0 to 1.8] | 0 [0.0 to 1.8]
  Fatigue: Any | 12.0 [7.8 to 17.3] | 12.0 [7.8 to 17.3]
  Fatigue: Mild | 7.5 [4.3 to 12.1] | 8.5 [5.0 to 13.3]
  Fatigue: Moderate | 4.0 [1.7 to 7.7] | 3.0 [1.1 to 6.4]
  Fatigue: Severe | 0.5 [0.0 to 2.8] | 0.5 [0.0 to 2.8]
  Headache: Any | 12.0 [7.8 to 17.3] | 11.5 [7.4 to 16.8]
  Headache: Mild | 9.5 [5.8 to 14.4] | 9.5 [5.8 to 14.4]
  Headache: Moderate | 2.0 [0.5 to 5.0] | 1.5 [0.3 to 4.3]
  Headache: Severe | 0.5 [0.0 to 2.8] | 0.5 [0.0 to 2.8]
  Joint pain: Any | 5.0 [2.4 to 9.0] | 4.0 [1.7 to 7.7]
  Joint pain: Mild | 3.0 [1.1 to 6.4] | 2.5 [0.8 to 5.7]
  Joint pain: Moderate | 2.0 [0.5 to 5.0] | 1.0 [0.1 to 3.6]
  Joint pain: Severe | 0 [0.0 to 1.8] | 0.5 [0.0 to 2.8]
  Muscle pain: Any | 14.5 [9.9 to 20.2] | 9.0 [5.4 to 13.9]
  Muscle pain: Mild | 10.0 [6.2 to 15.0] | 7.0 [3.9 to 11.5]
  Muscle pain: Moderate | 4.5 [2.1 to 8.4] | 1.5 [0.3 to 4.3]
  Muscle pain: Severe | 0 [0.0 to 1.8] | 0.5 [0.0 to 2.8]

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Vaccination to 1 Month After Vaccination
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were reported in this outcome measure. Exact 2-sided 95% confidence interval was based on the Clopper and Pearson method.
Time Frame: From vaccination on Day 1 up to 1 Month after vaccination
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: 18 to 49 Years | Cohort 2: >= 50 Years
Number analyzed (Participants) | 200 | 200
Percentage of participants | 1.5 [0.3 to 4.3] | 3.0 [1.1 to 6.4]

4. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) From Vaccination to 1 Month After Vaccination
Description: An SAE was any untoward medical occurrence at any dose that: resulted in death, was life threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, resulted in congenital anomaly/birth defect or was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic or that was considered to be an important medical event.
Time Frame: From vaccination on Day 1 up to 1 Month after vaccination
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Cohort 1: 18 to 49 Years | Cohort 2: >= 50 Years
Number analyzed (Participants) | 200 | 200
Percentage of participants | 0 | 0

5. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Pneumococcal Serotype-Specific Opsonophagocytic Activity (OPA) Titers From Before Vaccination to 1 Month After Vaccination
Description: GMFRs and 2-sided 95% confidence interval (CIs) were calculated by exponentiating the mean logarithm of fold rises and the corresponding CIs (based on the Student t distribution). Assay results below the lower limit of quantification (LLOQ) were set to 0.5*LLOQ in the analysis. Evaluable immunogenicity population: Eligible participants in the immunogenicity subset who received 1 dose of the intervention with at least 1 valid immunogenicity result from the blood sample collection within 27 to 49 days after vaccination, had no other major protocol deviations as determined by the clinician.
Time Frame: From before vaccination to 1 Month after vaccination
Population: Evaluable immunogenicity population evaluated. Number of participants analyzed= Number of participants in evaluable immunogenicity population. Number Analyzed = Number of evaluable participants with valid OPA titers for the specified serotype both before and after vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Cohort 1: 18 to 49 Years | Cohort 2: >= 50 Years
Number analyzed (Participants) | 50 | 49
Fold rise
  Serotype 1: number analyzed (Participants) | 47 | 41
  Serotype 1 | 24.3 [17.2 to 34.3] | 17.1 [10.9 to 26.9]
  Serotype 3: number analyzed (Participants) | 44 | 40
  Serotype 3 | 8.9 [5.7 to 13.8] | 8.8 [5.6 to 13.8]
  Serotype 4: number analyzed (Participants) | 43 | 42
  Serotype 4 | 15.2 [7.7 to 29.8] | 42.6 [22.0 to 82.6]
  Serotype 5: number analyzed (Participants) | 46 | 41
  Serotype 5 | 14.9 [8.6 to 25.8] | 24.3 [13.5 to 43.7]
  Serotype 6A: number analyzed (Participants) | 45 | 38
  Serotype 6A | 29.8 [16.3 to 54.5] | 30.9 [17.5 to 54.7]
  Serotype 6B: number analyzed (Participants) | 44 | 38
  Serotype 6B | 8.6 [5.0 to 15.0] | 11.6 [6.6 to 20.5]
  Serotype 7F: number analyzed (Participants) | 45 | 47
  Serotype 7F | 16.0 [9.2 to 27.9] | 24.1 [15.6 to 37.4]
  Serotype 9V: number analyzed (Participants) | 45 | 46
  Serotype 9V | 4.8 [3.2 to 7.1] | 9.5 [5.7 to 15.8]
  Serotype 14: number analyzed (Participants) | 46 | 40
  Serotype 14 | 5.8 [3.5 to 9.9] | 6.0 [3.3 to 10.9]
  Serotype 18C: number analyzed (Participants) | 44 | 46
  Serotype 18C | 21.4 [11.4 to 40.1] | 42.0 [22.4 to 78.6]
  Serotype 19A: number analyzed (Participants) | 46 | 42
  Serotype 19A | 15.0 [9.1 to 24.7] | 30.9 [18.1 to 52.6]
  Serotype 19F: number analyzed (Participants) | 44 | 39
  Serotype 19F | 13.1 [7.3 to 23.5] | 19.1 [10.5 to 35.0]
  Serotype 23F: number analyzed (Participants) | 46 | 47
  Serotype 23F | 46.2 [21.8 to 98.2] | 53.6 [28.3 to 101.4]
  Serotype 8: number analyzed (Participants) | 44 | 42
  Serotype 8 | 18.4 [10.5 to 32.4] | 38.2 [22.8 to 64.2]
  Serotype 10A: number analyzed (Participants) | 40 | 40
  Serotype 10A | 8.4 [5.0 to 14.0] | 31.1 [16.1 to 59.9]
  Serotype 11A: number analyzed (Participants) | 44 | 38
  Serotype 11A | 3.3 [2.3 to 4.7] | 9.5 [5.2 to 17.3]
  Serotype 12F: number analyzed (Participants) | 41 | 39
  Serotype 12F | 76.1 [33.4 to 173.7] | 75.2 [36.7 to 154.0]
  Serotype 15B: number analyzed (Participants) | 44 | 42
  Serotype 15B | 48.8 [22.2 to 107.0] | 86.2 [40.8 to 182.1]
  Serotype 22F: number analyzed (Participants) | 41 | 40
  Serotype 22F | 12.6 [7.8 to 20.4] | 30.8 [14.2 to 67.0]
  Serotype 33F: number analyzed (Participants) | 43 | 42
  Serotype 33F | 8.4 [5.0 to 14.0] | 11.7 [7.3 to 18.6]

ADVERSE EVENTS:
Time Frame: Systematic assessment: local reactions and systemic events recorded from Day 1 to Day 7 after vaccination; Non-systematic assessment: All-cause mortality, SAEs and other AEs recorded from day of vaccination (Day 1) up to 1 month after vaccination
Description: As all participants received 20vPnC the AEs section was reported together.
Groups:
- 20vPnC: Pneumococcal vaccine naive participants aged 18 to 49 years and >=50 years were administered 0.5 mL of 20vPnC vaccine, IM on Day 1 (Visit 1).
Arm/Group | 20vPnC
All-Cause Mortality (participants affected / at risk) | 0/400
Serious Adverse Events (participants affected / at risk) | 0/400
Other Adverse Events (participants affected / at risk) | 171/400
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 20vPnC (N=400)
Fatigue (FATIGUE) (General disorders) | 48
Injection site pain (PAIN) (General disorders) | 151
Injection site swelling (SWELLING) (General disorders) | 6
Pyrexia (FEVER) (General disorders) | 9
Arthralgia (JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 18
Myalgia (MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 47
Headache (HEADACHE) (Nervous system disorders) | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-12-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT05875727/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT05875727/SAP_001.pdf